CLINICAL TRIAL: NCT00851825
Title: The Effect of T-Tube and Pressure Support on Cardiorespiratory Variables and Heart Rate Variability During Weaning From Mechanical Ventilation
Brief Title: Heart Rate Variability During Weaning From Mechanical Ventilation
Status: Completed | Type: Observational
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Silvia Regina Rios Vieira, Hospital de Clinicas de Porto Alegre
Other Study IDs: 03-435
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2009-05-08 (Estimated); Status verified 2009-05

CONDITIONS: Critical Care; Weaning
Keywords: autonomic modulation; heart rate; pressure support ventilation; T-tube; Mechanical ventilation

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The discontinuation of mechanical ventilation (MV) and the recovery of spontaneous breathing can lead to important cardiovascular alterations due to changes in the intrathoracic pressure. The autonomic modulation assessed through heart rate variability (HRV) during weaning from MV and its impact on cardiorespiratory variables has not been well elucidated yet. To evaluate the effect of T-tube (TT) and pressure support ventilation (PSV) during weaning from MV on cardiorespiratory variables and heart rate variability.

DETAILED DESCRIPTION:
Thirty patients who had received MV for ≥ 48 hours and who met the criteria for weaning were assessed. Two different weaning methods were used and randomization was performed to choose one of the following sequences (baseline, PSV, rest, TT; or baseline, TT, rest, PSV). HRV was assessed by heart rate spectral analysis during MV, PSV, and TT. Each intervention lasted 30 minutes and there was a 30-minute rest period between the interventions. At the end of each period of time, the following cardiorespiratory variables were analyzed: respiratory rate (f), minute ventilation (VE), tidal volume (VT), rapid shallow breathing index (f/VT), peripheral oxygen saturation (SpO2), heart rate (HR) and blood pressure. In the HRV, the total spectral power (TP), the low frequency (LF) and the high frequency (HF) components, and the ratio between the low/high frequency (LF/HF) components were calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with respiratory failure receiving MV for more than 48 hours
* for weaning from MV according to the parameters previously defined were selected to participate in this study

Exclusion Criteria:

* arterial hypotension (systolic blood pressure < 100mmHg), severe brain disease, barotraumas, presence of thoracic drain or tracheostomy, using vasoactive and sedative drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with respiratory failure receiving MV for more than 48 hours, who had been admitted to the Intensive Care Unit (ICU) of the Hospital de Clínicas de Porto Alegre, and who met the criteria for weaning from MV according to the parameters previously defined were selected to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2003-03; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
heart rate variability analysis | minutes

SECONDARY OUTCOMES:
Cardiorespiratory variables | minutes

CONTACTS AND LOCATIONS:
Overall Officials: Silvia R Veira, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil